CLINICAL TRIAL: NCT05315115
Title: To Investigate the Effects of Four Weeks of Intensive Chiropractic Care When Added to Usual Care for Adults With Spinal Cord Injuries.
Brief Title: Effects of Intensive Chiropractic Care to Usual Care for Adults With Spinal Cord Injuries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/01287 Imran Amjad
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Research
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A registered chiropractor will assess the entire spine, and both sacroiliac joints will be assessed for vertebral subluxation by a registered chiropractor. The clinical indicators that will be used to assess the function of the spine before spinal adjustment intervention include assessing for joint tenderness to palpation manually palpating for a restricted intersegmental range of motion, assessing for palpable asymmetric intervertebral muscle tension, and any abnormal or blocked joint play and end-feel of the joints.
  Interventions: Other: Chiropractic Care; Other: Physical therapy intervention
- Control group (Sham Comparator): The participant's head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor.No spinal adjustment will be performed during any control intervention.
  Interventions: Other: Sham intervention; Other: Physical therapy intervention

INTERVENTIONS:
Other: Sham intervention — The participant's head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor. The sham intervention will also include the participants moving into adjustment setup positions similar to how the chiropractor would typically set up a patient with no joint pre-loading or adjustive thrust.
  Arms: Control group
Other: Chiropractic Care — A registered chiropractor will assess the entire spine, and both sacroiliac joints will be assessed for vertebral subluxation by a registered chiropractor. The clinical indicators that will be used to assess the function of the spine before spinal adjustment intervention include assessing for joint tenderness to palpation manually palpating for a restricted intersegmental range of motion, assessing for palpable asymmetric intervertebral muscle tension, and any abnormal or blocked joint play and end-feel of the joints.
  Arms: Experimental group
Other: Physical therapy intervention — The standardized treatment protocol will be provided according to the guidelines, which will include various modalities and treatment approaches, including stretching exercises; massage; strengthening exercises of weak muscles, weight-bearing, balance (static and dynamic) and gait training; electrical stimulation; treadmill use; and endurance training for the improvement of gait, motor function, strength and functional mobility in Spinal Cord Injuries children, where Conventional Therapy will be provided according to the respective needs of the individual patient.

SUMMARY:
To determine the effects of chiropractic care on spasticity, functional outcomes and quality of life in Spinal Cord Injuries in adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults with both genders (Male and Female).
* Age above 20 years.
* Spinal Cord Injuries adults.

Exclusion criteria

* Spinal Cord Injury due to Traumatic Brain Injury.
* Patients having cognitive impairments.
* Patients having associated Neurological Pathologies.
* Patients who are unable to follow the treatment plan.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | Baseline
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability for a variety of populations and is not specific to any diagnosis. FIM is comprised of 18 items, grouped into 2 subscales - motor and cognition. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item. This tool will be measured at baseline.
Functional Independence Measure (FIM) | 4 weeks
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability for a variety of populations and is not specific to any diagnosis. FIM is comprised of 18 items, grouped into 2 subscales - motor and cognition. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item. This tool will be measured after 4 weeks.
ASIA scale | Baseline
  The American Spinal Injury Association (ASIA) impairment scale describes a person's functional impairment as a result of a Spinal Cord Injury. This scale indicates how much sensation a person feels after light touch and a pinprick at multiple points on the body and tests key motions on both sides of the body. This tool will be measured at baseline.
ASIA scale | 4 weeks
  The American Spinal Injury Association (ASIA) impairment scale describes a person's functional impairment as a result of a Spinal Cord Injury. This scale indicates how much sensation a person feels after light touch and a pinprick at multiple points on the body and tests key motions on both sides of the body. This tool will be measured after 4 weeks.
Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire (SSSMQ) | Baseline
  The SSSMQ is a newly developed tool to assess Spine Dysfunction Characteristics, logical and Psychological Stress Symptoms, and Multimodal and Sensorimotor Integration Dysfunction Symptoms. A baseline assessment of a participant will be done before the start of the intervention.
Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire (SSSMQ) | 4 weeks
  The SSSMQ is a newly developed tool to assess Spine Dysfunction Characteristics, logical and Psychological Stress Symptoms, and Multimodal and Sensorimotor Integration Dysfunction Symptoms. A baseline assessment of a participant will be done before the start of the intervention. This tool will be measured after 4 weeks.
36-Item Short Form Survey (SF-36) | Baseline
  The SF-36 was originally designed as a generic health measure but has also been applied to specific disease populations. It comprises 36 questions that cover eight domains of health. Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to the high quality of life. A baseline assessment of a participant will be done before the start of the intervention.
36-Item Short Form Survey (SF-36) | 4 weeks
  The SF-36 was originally designed as a generic health measure but has also been applied to specific disease populations. It comprises 36 questions that cover eight domains of health. Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to the high quality of life. This tool will be measured after 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: IMRAN AMJAD, PhD, Principal Investigator — Riphah International University
Locations (1):
- National Institute of rehabilitation medicine., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No